CLINICAL TRIAL: NCT01300650
Title: Pilot Study of the Safety and Efficacy of Anakinra (Recombinant Human Interleukin-1 Receptor Antagonist) in Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIR-HF Pilot Study; 1KL2RR031989-01 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
Keywords: Heart failure; Inflammation; Interleukin-1; Cardiopulmonary exercise
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anakinra (Experimental)
  Interventions: Drug: Anakinra

INTERVENTIONS:
Drug: Anakinra — Anakinra 100 mg subcutaneous injection daily

SUMMARY:
This is an open-label, non-randomized, pilot-study to evaluate the effect of Interleukin-1 blockade on exercise capacity in patients with heart failure. Subjects will undergo cardiopulmonary exercise testing at baseline and after 2-weeks treatment with anakinra (recombinant human Interleukin-1 receptor antagonist).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of heart failure
* Recent echocardiogram documenting left ventricular ejection fraction <40%
* High sensitivity C-reactive protein >2 mg/L.

Exclusion Criteria:

* Recent changes (previous 3 months) in HF maintenance medications (beta-blockers, angiotensin converting enzyme [ACE] inhibitors, aldosterone antagonists, vasodilators, cardiac glycosides, diuretics)
* Hospitalization for worsening HF or acute decompensated HF within the previous 12 months
* Anticipated need for cardiac resynchronization therapy (CRT) or automated-implantable cardioverter defibrillator (AICD)
* Angina or electrocardiograph (ECG) changes that limit maximum exertion during cardiopulmonary exercise testing or baseline ECG changes that limit the ability to detect ischemia (i.e. left bundle-branch block).
* Recent (<14 days) use of anti-inflammatory drugs (not including NSAIDs), chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus), malignancy, active infection, or any comorbidity limiting survival or ability to complete the study
* Severe kidney dysfunction (eGFR <30 mL/min)
* Coagulopathy (INR >1.5), thrombocytopenia (<50,000/mm3), or leukopenia (absolute neutrophil count <1,500/mm3)
* Pregnancy (female patients will be required to take a urine pregnancy test)
* Latex or rubber allergy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Van Tassell BW, Arena RA, Toldo S, Mezzaroma E, Azam T, Seropian IM, Shah K, Canada J, Voelkel NF, Dinarello CA, Abbate A. Enhanced interleukin-1 activity contributes to exercise intolerance in patients with systolic heart failure. PLoS One. 2012;7(3):e33438. doi: 10.1371/journal.pone.0033438. Epub 2012 Mar 16. PMID 22438931

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients had elevated hsCRP (>2 mg/L) and were enrolled in the study.
Pre-assignment Details: 2 patients withdrew consent prior to beginning the study. 1 patient underwent a change in heart failure medication prior to beginning the study and was therefore withdrawn from the study. The 8 remaining patients began the study interventions.
Groups:
- Anakinra: Anakinra 100 mg subcutaneous daily injection
Period: Overall Study
Arm/Group | Anakinra
Started | 8
Completed | 7
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anakinra
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Median Interval Change From Baseline in Peak VO2
Description: Peak VO2 is a measurement of oxygen consumption rate during exercise (milliliters of oxygen per minute). It is calculated by continuous measurement of oxygen consumed during exercise while patients breath through a mask/tube. To account for variability in patient size, the oxygen consumption is divided by patient body weight.
  The outcome measure time frame was 14 days. This means that change in peak VO2 was calculated as the difference between peak VO2 at baseline and 14 days. To calculate this change, we used the mathematical process of subtraction (change in peak VO2 = Peak VO2 [day 14] - Peak VO2 [baseline])
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Anakinra
Number analyzed (Participants) | 7
mL/kg/min | 3.90 [2.30 to 4.95]

2. Primary Outcome: Median Interval Change From Baseline in the Minute Ventilation and Carbon Dioxide Production (VE/VCO2 Slope)
Description: The VE/VCO2 slope is calculated as the ratio of minute ventilation (VE) and carbon dioxide production (VCO2). Because these measurements share the same units, the resultant ratio is unitless.
  Change in VE/VCO2 slope was calculated as the change in VE/VCO2 slope between baseline and 14 days. We therefore calculated the difference between VE/VCO2 slope measurements that occurred at baseline and at 14 days (change in VE/VCO2 slope = VE/VCO2 slope [day 14] - VE/VCO2 slope [baseline])
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: (unitless)
Arm/Group | Anakinra
Number analyzed (Participants) | 7
(unitless) | -2.10 [-4.10 to -0.55]

3. Secondary Outcome: Interval Change From Baseline in Heart Failure Symptoms as Measured by Duke Activity Status Index (DASI)
Description: The Duke Activity Status Index (DASI) is a scale that quantifies patients' ability to perform various tasks. The scale ranges from 0 (unable to perform any tasks) to 58.20 (able to perform all tasks). Higher scores reflect improved activity or improved heart failure symptoms. Lower scores reflect worsened ability or worsened heart failure symptoms.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Anakinra: Anakinra 100 mg subcutaneous injection
Arm/Group | Anakinra
Number analyzed (Participants) | 7
units on a scale | 6 [0 to 20.2]

4. Other Pre Specified Outcome: Interval Change From Baseline in Biomarkers (High-sensitivity C-reactive Protein, Whole Blood Assay, Brain Natriuretic Peptide)
Time Frame: 14 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Correlation Between Interval Changes in Biomarkers, Peak VO2, and VE/VCO2
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Anakinra
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anakinra (N=8)
Flu-like symptoms (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No